CLINICAL TRIAL: NCT01552434
Title: A Phase I Trial of Bevacizumab, Temsirolimus Alone and in Combination With Valproic Acid, or Cetuximab in Patients With Advanced Malignancy and Other Indications
Brief Title: Bevacizumab and Temsirolimus Alone or in Combination With Valproic Acid or Cetuximab in Treating Patients With Advanced or Metastatic Malignancy or Other Benign Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0061; NCI-2012-00347 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0061 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-03-07; First posted 2012-03-13 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Neoplasm; Castleman Disease; Digestive System Carcinoma; Erdheim-Chester Disease; Lip and Oral Cavity Carcinoma; Lymphangioleiomyomatosis; Malignant Endocrine Neoplasm; Malignant Female Reproductive System Neoplasm; Malignant Male Reproductive System Neoplasm; Malignant Neoplasm; Malignant Respiratory Tract Neoplasm; Malignant Thoracic Neoplasm; Malignant Urinary System Neoplasm; Mesothelial Neoplasm; Metastatic Malignant Neoplasm; Metastatic Urothelial Carcinoma; Neurofibromatosis Type 2; Recurrent Adult Soft Tissue Sarcoma; Recurrent Breast Carcinoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Digestive System Carcinoma; Recurrent Female Reproductive System Carcinoma; Recurrent Male Reproductive System Carcinoma; Recurrent Malignant Neoplasm; Recurrent Pharyngeal Carcinoma; Recurrent Thyroid Gland Carcinoma; Refractory Malignant Neoplasm; Soft Tissue Neoplasm; Stage III Breast Cancer AJCC v7; Stage III Pharyngeal Cancer; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7; Stage IV Pharyngeal Cancer; Stage IVA Pharyngeal Cancer; Stage IVB Pharyngeal Cancer; Stage IVC Pharyngeal Cancer; Thyroid Gland Neoplasm
Keywords: Temsirolimus; CCI-779; Torisel; Bevacizumab; Avastin; rhuMAb-VEGF; Anti-VEGF Monoclonal Antibody; Advanced Cancers; Advanced Malignancy; Metastatic; cancer; Cetuximab; C225; Erbitux; IMC-C225; Valproic Acid
MeSH Terms: conditions — Castleman Disease; Erdheim-Chester Disease; Mouth Neoplasms; Lymphangioleiomyomatosis; Endocrine Gland Neoplasms; Neoplasms; Urologic Neoplasms; Neoplasms, Mesothelial; Neoplasm Metastasis; Carcinoma, Transitional Cell; Neurofibromatosis 2; Sarcoma; Breast Neoplasms; Recurrence; Pharyngeal Neoplasms; Thyroid Neoplasms; Soft Tissue Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Cetuximab; temsirolimus; Sirolimus; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group I (temsirolimus, bevacizumab, cetuximab) (Experimental): Patients receive temsirolimus IV over 30-60 minutes on days 1, 8, 15, and 22; bevacizumab IV over 30-90 minutes on days 1 and 15; and cetuximab IV over 60-120 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Biological: Cetuximab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temsirolimus
- Group II (temsirolimus, bevacizumab, valproic acid) (Experimental): Patients receive temsirolimus and bevacizumab as in Group I and valproic acid PO on days 1-7 and 15-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temsirolimus; Drug: Valproic Acid
- Group III (temsirolimus, bevacizumab) (Experimental): Patients receive temsirolimus and bevacizumab as in Group I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temsirolimus

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Biological: Cetuximab — Given IV
  Other Names: Cetuximab Biosimilar CMAB009; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Group I (temsirolimus, bevacizumab, cetuximab)
Other: Laboratory Biomarker Analysis — Optional correlative studies
Other: Pharmacological Study — Optional correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
Drug: Valproic Acid — Given PO
  Other Names: Depakene; Stavzor; Valproate
  Arms: Group II (temsirolimus, bevacizumab, valproic acid)

SUMMARY:
This phase I trial studies the side effects and best dose of bevacizumab and temsirolimus alone or in combination with valproic acid or cetuximab in treating patients with a malignancy that has spread to other places in the body or other disease that is not cancerous. Immunotherapy with bevacizumab and cetuximab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as valproic acid, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether bevacizumab and temsirolimus work better when given alone or with valproic acid or cetuximab in treating patients with a malignancy or other disease that is not cancerous.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated doses (MTDs) and dose-limiting toxicities (DLTs) of treatment with bevacizumab and temsirolimus in combination and plus valproic acid or cetuximab.

SECONDARY OBJECTIVES:

I. Preliminary descriptive assessment of anti-tumor efficacy of each combination.

II. Preliminary assessment of the pharmacokinetic, pharmacodynamic markers of target inhibition and correlates of response (optional).

OUTLINE: This is a dose-escalation study of bevacizumab and temsirolimus. Patients are assigned to 1 of 3 treatment groups.

GROUP I: Patients receive temsirolimus intravenously (IV) over 30-60 minutes on days 1, 8, 15, and 22; bevacizumab IV over 30-90 minutes on days 1 and 15; and cetuximab IV over 1-2 hours on days 1, 8, 15, and 22.

GROUP II: Patients receive temsirolimus and bevacizumab as in Group I and valproic acid orally (PO) daily on days 1-7 and 15-21.

GROUP III: Patients receive temsirolimus and bevacizumab as in Group I.

In all groups, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or have no standard therapy that induces a complete response of at least 10% or improves survival by at least three months; in addition, patients with disease that are "benign" by pathology, but relentlessly progressive, leading to disability, pain, and premature death in the majority of cases (including, but not limited to lymphangioleiomyomatosis [LAM], type 2 neurofibromatosis [NF], Erdheim Chester disease, and Castleman's disease) may also be considered for enrollment
* Patients should be at least four weeks from the last day of therapeutic radiation or cytotoxic chemotherapy or from antibody therapy, or at least five half-lives from non-cytotoxic targeted or biologic therapy; patients may have received palliative radiation immediately before (or during) treatment provided radiation is not to the only target lesion available
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Karnofsky >= 60%
* Lansky performance status of >= 60% for participants 16 years old or younger
* Absolute neutrophil count >= 1,000/mL
* Platelets >= 50,000/mL
* Creatinine =< 3 X upper limit of normal (ULN)
* Total bilirubin =< 3.0
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 X ULN
* Fasting level of total cholesterol of no more than 350 mg/dL
* Triglyceride level of no more than 400 mg/dL
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days after the last dose
* Ability to understand and the willingness to sign a written informed consent document
* Patients may not be receiving any other investigational agents and/or any other concurrent anticancer agents or therapies

Exclusion Criteria:

* Patients with clinically significant unexplained bleeding within 28 days prior to entering the study
* Uncontrolled systemic vascular hypertension (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg on medication)
* Patients with clinically significant cardiovascular disease: History of CVA (cerebrovascular accident) within 6 months, myocardial infarction or unstable angina within 6 months, unstable angina pectoris
* Pregnant or breast-feeding women
* History of hypersensitivity to bevacizumab, murine products, or any component of the formulation
* History of hypersensitivity to temsirolimus or its metabolites (including sirolimus), polysorbate 80, or to any component of the formulation
* History of hypersensitivity to cetuximab, murine products, or any component of the formulation
* Patients that are taking cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inducers and/or inhibitors; if a patient has a history of taking CYP3A4 inducers and/or inhibitors prior to enrollment on the protocol, it is strongly recommended that the patient stops the drug and waits at least 5 half-lives of said drug before initiating therapy on protocol
* Colorectal cancer patients with known v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS) mutation (for the arm combining bevacizumab, temsirolimus and cetuximab)
* Patients who have had major surgery within 6 weeks of enrollment in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2012-03-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of bevacizumab, defined as the dose level below the dose at which 2 of 6 patients experience drug-related dose limiting toxicity (DLT) | 4 weeks
  Graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
MTD of temsirolimus, defined as the dose level below the dose at which 2 of 6 patients experience DLT | 4 weeks
  Graded by the NCI CTCAE version 3.0.

SECONDARY OUTCOMES:
Anti-tumor efficacy of each combination (objective response) | Up to 6 years
  Will be determined by Response Evaluation Criteria In Solid Tumors and World Health Organization criteria
Levels of surrogate anti-angiogenesis markers | Up to week 4 of course 1
  Correlated with anti-tumor activity.

OTHER OUTCOMES:
The properties of the tissue microvasculature. | Up to week 4 of course 1
  The properties of the tissue microvasculature measured by Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) include parameters:
  volume transfer coefficient, (Ktrans), fractional volume (ve), and rate constant (kep).For each of these parameters, an exploratory analysis of change from baseline will be conducted which will include mean, median, standard deviation, and 95% confidence limits.

CONTACTS AND LOCATIONS:
Overall Officials: Sarina A Piha-Paul, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Piha-Paul SA, Tseng C, Thompson E, Stafford RJ, Le H, Kang L, Fu S, Tsimberidou A, Blumenschein G Jr, Ahnert JR, Slopis JM, Hong D, Niang A, Meric-Bernstam F, Ng CS, Westin S, Sood AK. Phase I Study of Bevacizumab and Temsirolimus Combination Therapy in Advanced Malignancies: Safety, Efficacy, and Ovarian Cancer Expansion. Oncologist. 2025 Dec 13:oyaf413. doi: 10.1093/oncolo/oyaf413. Online ahead of print. PMID 41389341
- [Derived] Nelson BE, Tsimberidou AM, Fu X, Fu S, Subbiah V, Sood AK, Rodon J, Karp DD, Blumenschein G, Kopetz S, Pant S, Piha-Paul SA. A Phase I Trial of Bevacizumab and Temsirolimus in Combination With Valproic Acid in Advanced Solid Tumors. Oncologist. 2023 Dec 11;28(12):1100-e1292. doi: 10.1093/oncolo/oyad158. PMID 37311055
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org